CLINICAL TRIAL: NCT00202150
Title: Primary Care Management/Action Plans for Advanced Chronic Diseases (The RoadMAP Project)
Brief Title: Primary Care Management/Action Plans for Advanced Chronic Diseases
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G03-02765
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure; Chronic Obstructive Lung Disease
Keywords: Advanced chronic diseases; Heart failure; Chronic obstructive lung disease; primary care; Chronic Care
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Behavioral: Application of a management action plan

SUMMARY:
Patients living with advanced chronic diseases (ACD), such as congestive heart failure (CHF) and chronic obstructive lung disease (COPD) present substantial care and economic challenges for the health care system due to frequent emergency room visits and acute care hospitalizations. Morbidity and mortality is high in these complex populations, and patient quality of life is often compromised.

Care of patients with ACD occurs across health care sectors, by providers in the acute, primary and community settings. Despite recent efforts to enhance the care of patients with ACD, through multidisciplinary disease management programs, variations and gaps exist along the continuum of care. The available evidence suggests that there are opportunities to optimize the primary care of patients with ACD. We are proposing to build upon the current evidence and guidelines for disease management programs, our existing specialized resources, our existing primary care practices, and develop and test a model of care that is primary care based, sensitive to the unique demands and characteristics of different primary practices. Our goal is to design linkages and care strategies of relevance and importance to the primary care providers who care for patients with advanced COPD and CHF.

This demonstration project is a randomized controlled clinical trial of the RoadMAP program (intervention) delivered by a Primary Care Nurse Specialist (PCNS) compared to usual care (control group). The primary outcomes will be degree of adherence to clinical practice guidelines. Secondary outcomes will be patient satisfaction, quality of life, use of community-based services, number of emergency room visits, and number of hospitalizations.

DETAILED DESCRIPTION:
The available evidence suggests that there are opportunities to optimize the primary care of patients with ACD. We are proposing to build upon the current evidence and guidelines for disease management programs, our existing specialized resources, our existing primary care practices, and develop and test a model of care that is primary care based, sensitive to the unique demands and characteristics of different primary practices. Our goal is to design linkage and care strategies of relevance and importance to the primary care providers who care for patients with advanced COPD and CHF.

The study is a randomized controlled clinical trial of the RoadMAP program (intervention) delivered by a PCNS compared to usual care (control group). The primary outcome will be degree of adherence to clinical practice guidelines. Secondary outcomes will be patient satisfaction, quality of life, use of community-based services, number of emergency room visits, and number of hospitalizations. The purpose of the RoadMAP program is to improve the care of people with advanced stage COPD and CHF. Specifically, activities will be aimed at improving patients' self care ability, facilitating access to the most appropriate services, ensuring medical treatment according to consensus guidelines and promoting consistency of health care communication. Adherence to guidelines is a process that involves activities by the patient, PCNS, and the Primary Care Physician. The PCNS would follow-up the patient again at approximately one month after initial contact and then every 3 months, to assess and monitor adherence to the proposed MAP by the patient, the physician, and the nurse. Patients will have the option of returning to the physician office or to be monitored by phone. An office visit will be recommended if there is a perceived need for medical assessment and intervention. The family physician would continue to see the patient as required in order to carry out the medical portion of the MAP and to deal with other primary care problems as needed. Additionally, the PCNS would be available to work with nurses and other health professionals in each primary care practice in the provision of care to the ACD patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Chronic Heart Failure
* diagnosis of Chronic Obstructive Pulmonary Disease

Exclusion Criteria:

* living in a nursing home
* inability to give informed consent
* involved in other studies of CHF or COPD

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2004-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Degree of adherence to the clinical practice guidelines.

SECONDARY OUTCOMES:
Patient satisfaction
General health related quality of life
Therapeutic Self Care
Number of referrals to community-based services
Number of emergency room visits annually
Number of hospitalizations annually

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Godwin, MD MSc, Principal Investigator — Centre for Studies in Primary Care; Joan Tranmer, RN PhD, Principal Investigator — Kingston Health Sciences Centre
Locations (1):
- Centre for Studies in Primary Care, Kingston, Ontario, Canada